CLINICAL TRIAL: NCT04005417
Title: Bioavailable Stannous Fluoride Dentifrice Meta-Analyses: Effects on Dentine Hypersensitivity and Enamel Erosion
Brief Title: Meta-analysis of Stannous Fluoride Dentifrice and the Effects on Dentine Hypersensitivity
Status: Completed | Type: Observational
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019SnF2SensitivityAnalysis
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stannous fluoride dentifrice: Twice daily brushing
  Interventions: Drug: Stannous fluoride dentifrice
- Positive control dentifrice: Twice daily brushing
  Interventions: Drug: Positive control dentifrice
- Negative control dentifrice: Twice daily brushing
  Interventions: Drug: Negative control dentifrice

INTERVENTIONS:
Drug: Stannous fluoride dentifrice — Stannous fluoride (0.454%) dentifrice
  Groups: Stannous fluoride dentifrice
Drug: Positive control dentifrice — Positive control dentifrice containing potassium nitrate or arginine.
  Groups: Positive control dentifrice
Drug: Negative control dentifrice — Negative control dentifrice containing either sodium fluoride (0.243%) or sodium monofluorophosphate (0.76%)
  Groups: Negative control dentifrice

SUMMARY:
The aim of this 11 study analysis was to compare the effect of bioavailable stannous fluoride (SnF2) on dentine hypersensitivity versus a positive or negative control dentifrice.

ELIGIBILITY:
Subjects were excluded from this study for the following reasons;

* severe periodontitis
* at discretionary of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This meta-analysis includes healthy adult male and females.
Sampling Method: Probability Sample
Enrollment: 1036 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Air Challenge | Up to 8 weeks
  The Schiff Sensitivity Scale is assessed for each test tooth via an evaporative air challenge. The examiner records the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth.
Change from Baseline in Tactile Threshold | Up to 8 weeks
  Tactile Threshold is measured using a Yeaple probe. Testing is performed beginning at 10 g. The examiner records tactile scores for responding teeth. After treatment, testing begins at 10 g and increases by 10 g to a maximum of 50 g. The higher the tactile threshold, the less sensitive the tooth. Each successive challenge increases until a "yes" response is repeated. If a second "yes" is not obtained, the force setting is increased to the next step and continued until a force is found which elicits two consecutive "yes" responses and is recorded as the threshold on the Tactile Sensitivity Score form.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple P&G Investigation Clinical Sites, Cincinnati, Ohio, United States